CLINICAL TRIAL: NCT05601635
Title: A Pilot Study to Demonstrate Butyrate Generation in Stool in Response to Oral Administration of ButyraGen™ in Healthy Human Subjects
Brief Title: ButyraGen™, Short Chain Fatty Acids and Gut Microbiome
Acronym: BG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-2023-25
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose (Active Comparator): Dietary supplement containing 200 mg of active ingredient tributyrin
  Interventions: Dietary Supplement: ButyraGen™
- Low dose (Active Comparator): Dietary supplement containing 100 mg of active ingredient tributyrin
  Interventions: Dietary Supplement: ButyraGen™

INTERVENTIONS:
Dietary Supplement: ButyraGen™ — ButyraGen™ contains tributyrin as the primary active as well as Sunfiber®, a partially hydrolyzed guar fiber, and acacia fiber.

SUMMARY:
This study is being conducted to demonstrate short chain fatty acid (SCFA), specifically butyrate, generation in stool, blood and urine in response to oral intake of ButyraGen™.

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening.

This is a single-center study will follow a randomized, single-blinded parallel design with two doses. It features a 1-week intake of control followed by 3 weeks of either low dose (200 mg ButyraGen, containing 100 mg tributyrin) or high dose (400 mg, containing 200 mg tributyrin) of intervention to evaluate the effects of the active ingredient tributyrin after chronic intake in generally healthy individuals.

A planned sample size of 24 will be enrolled in the study. This study will require one initial screening visit, a pre-study visit, and 6 study day visits. The study will last about 5 weeks to complete all study procedures for each participant.

The initial screening visit will provide subjects with their site-specific, IRB approved informed consent document prior to the start of any study-related procedures. Subject eligibility will be determined through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), fasting blood sample screened for complete blood count (CBC) and basic metabolic panel (BMP), and surveys related to general eating, health, mood and exercise habits.

Subjects will be randomized to 1 of 2 interventions: low dose (100 mg - tributyrin) or high does (200 mg - tributyrin). All subjects will receive 1 week of control (0 mg - tributyrin), then same treatment (low or high dose) for the remaining duration of the study. Treatment codes will be maintained by the principal investigator. Two of the 6 study days (first and last) will last ~7 hours and include a lactulose-mannitol test. In general, this test will ask you to collect your 1st urine of the day, drink a sugary beverage and collect all urine for the next 6 hours after the drink. The other 4 study days will last ~2 hours. Subjects will be required to remain at the Clinical Nutrition Research Center for the duration of the visit. Fasting blood samples will be collected via a butterfly needle by a certified phlebotomist.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female, 18 years of age, inclusive.
* Subject has a BMI of 20.0-30.0 kg/m2, inclusive and a weight ≥ 110 lb. at the screening visit.
* Subject is willing to maintain his/her usual physical activity pattern throughout the study period.
* Subject is willing to follow study instructions, including compliance with certain dietary restrictions, consumption of study products, and study visit schedule.
* Subject is judged to be in good health on the basis of the medical history.
* Subject is willing to abstain from alcohol consumption for 24 hours prior to the study visit.
* Subject is willing to maintain a stable dose of current medications not interfering with study outcomes, including birth control, throughout the study duration.
* Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator/s and is willing to complete study procedures.

Exclusion Criteria:

* Subject has fasting finger prick glucose >125 mg/dL.
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at the screening visit.
* Subject has had major trauma or a surgical event within 2 months of study visit 1.
* Subject has had a weight change ≥4.5 kg within 2 months of visit, taking weight loss drugs, or has had bariatric surgery or other weight reduction surgery (ie. liposuction, laser fat removal, etc)
* Subject has a history or presence of clinically important endocrine, cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary, or gastrointestinal disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
* Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Subject has a history of extreme dietary habits, as judged by the Investigator (e.g., Atkins diet, etc.).
* Subject has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
* Subject has a known intolerance or sensitivity to any ingredients in the study products.
* Subject has used medications known to influence carbohydrate and lipid metabolism, including, but not limited to adrenergic blockers, diuretics, hypoglycemic medications, and systemic corticosteroids 2 weeks prior to visit 0 and throughout the study or other medication(s) that may interfere with results of study.
* Subject taking fiber supplements.
* Subject taking systemic steroids, extreme alcohol use, or drug user.
* Subject has a vein access score of less than 7
* Subject is a female who is pregnant, planning to be pregnant during the study period or lactating.
* Subject is a current smoker. Past smoker abstinence for less than 1 years.
* Subject has participated in any clinical trial within 30 days prior to enrollment unless otherwise approved by the study Investigator.
* Subjects who are vegan or vegetarian
* Subjects who work overnight shift (e.g 3rd shift)
* Subject who donated blood within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
SCFAs in stool, blood and urine samples | Baseline to 4 weeks
  Outcome measure will be quantified via GC-FID

SECONDARY OUTCOMES:
Lactulose-mannitol test for leaky gut | Baseline to 4 weeks
  Outcome measure will be analyzed by Genova Diagnostics
Questionnaire for study product tolerability | Baseline to 4 weeks
  Yes or no question for experiences felt during study. If yes, rated based on how often - "much less than usual" to "much more than usual".

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No